CLINICAL TRIAL: NCT04370600
Title: A Phase 1, Crossover, Pharmacokinetic Study of Nutritional Ketosis on Exercise Capacity, Metabolic Adaptations, and Myocardial Function in Chronic Ambulatory Heart Failure
Brief Title: Nutritional Ketosis in Heart Failure
Acronym: INNKA-HF
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: JT#15471
Record Dates: First submitted 2020-03-10; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Chronic Heart Failure
Keywords: ketosis; beta-hydroxybutyrate; insulin; bioenergetics; exercise tolerance; metabolic; diabetes
MeSH Terms: conditions — Ketosis; Insulin Resistance; Diabetes Mellitus | interventions — 3-Hydroxybutyric Acid; Esters

STUDY DESIGN:
Intervention Model Description: Biological drug + placebo (Group A) or placebo + biological drug (Group B)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): These patients will receive ketone supplementation between visits 1 and 2 and will receive placebo drink between visits 2 and 3 (after the washout period).
  Interventions: Drug: beta hydroxybutyrate (BHB) ester; Drug: Placebo
- Group B (Active Comparator): These patients will receive ketone supplementation between visits 2 and 3 (after the washout period) and will receive placebo drink between visits 1 and 2
  Interventions: Drug: beta hydroxybutyrate (BHB) ester; Drug: Placebo

INTERVENTIONS:
Drug: beta hydroxybutyrate (BHB) ester — Ketone supplementation given 3x/day (60mL per dose, or 22g BHB)
  Other Names: Delta G
Drug: Placebo — Denatonium benzoate + HVMN ketone placebo flavor mix + Stevia

SUMMARY:
Chronic, ambulatory heart failure patients will be given ketone ester dietary supplementation to determine therapeutic efficacy, metabolic adaptation, pharmacokinetics, associated cognitive changes, and safety within this patient cohort in order to establish preliminary data to later conduct a multi-center randomized clinical trial.

DETAILED DESCRIPTION:
We previously demonstrated a metabolic signature of increased ketone utilization-increased peripheral blood concentration of beta-hydroxybutyrate (BHB) and decreased myocardial concentration of BHB-and markedly decreased acylcarnitine levels in the failing human myocardium procured from lean, non-diabetic patients with advanced heart failure at the time of cardiac transplantation. In this working model of the metabolic adaptations in human heart failure where the mobilization of lipids and ketones are required for an energetically deficient, failing heart it is likely that the development of insulin resistance may be adaptive since increased insulin or insulin signaling would put a brake on the hydrolysis of lipids and hepatic ketogenesis. In parallel with the recent discovery that the failing human heart is reliant on ketones, investigators at Oxford and the NIH have identified a nutritional ketone supplement that reliably increases the serum concentration of BHB in humans.

We hypothesize that the induction of ketosis by exogenous administration of the nutritional ketone monoester will improve myocardial function in heart failure by increasing the energetic substrate available to the myocardium, in essence supporting the energetic deficit of the failing human heart which we have demonstrated to be reliant on ketone bodies for fuel given the limited myocardial oxidation of glucose.

This is a prospective, double-blinded, sequence control crossover trial enrolling NYHA Class II-III ambulatory heart failure patients to receive either ketone mono-ester drink versus placebo for two weeks. Following 2 weeks of therapy, echocardiogram and peak exercise test will be performed. There will be a 1-week "washout" period between phases. Subjects will serve as their own controls for this crossover study, as each will have both baseline testing and testing in the setting of mild nutritional ketosis.

ELIGIBILITY:
Inclusion Criteria:

1. Equal to or greater than 18 years of age
2. Diagnosis of heart failure and be classified as NYHA Class II or III either pre-enrollment or at the time of enrollment
3. Stable medical therapy for at least 1 month prior to enrollment
4. Taking appropriate daily cardiac medications as determined by the principal investigator, who is a heart failure specialist

Exclusion Criteria:

1. Atrial fibrillation
2. Inability to exercise on a supine bicycle.
3. Moderate or greater valvular disease.
4. Hemoglobin <10 g/dL.
5. Daily insulin use
6. Hypertrophic, infiltrative, or inflammatory cardiomyopathy.
7. Pericardial disease.
8. Current angina due to clinically significant obstructive epicardial coronary disease
9. Acute coronary syndrome or coronary intervention within the past 2 months.
10. Primary pulmonary arteriopathy.
11. Known clinically significant lung disease defined as:

    1. Current use of supplemental oxygen, aside from nocturnal O2 for the treatment of obstructive sleep apnea
    2. The use of steroids/antibiotics within the past 6 months for an acute exacerbation of obstructive pulmonary disease
    3. Most proximal pulmonary function test indicating severe obstructive disease, defined as an FEV1<50% predicted in the context of an FEV1/FVC ratio of <0.70 ("Stage III COPD according to GOLD Criteria). (note: only to be used if the subject had PFTs prior to screening)
    4. Most proximal 6-minute walk test during which the subject experienced arterial desaturation (<94%) without a subsequent normal study.
12. Ischemia on stress testing without subsequent revascularization or left heart catheterization showing non-obstructive epicardial coronary disease.
13. Significant liver disease impacting synthetic function or volume control.
14. Uncontrolled hypertension: BP >180/110 at baseline.
15. eGFR <30 mL/min/m2 or Cr >2.5.
16. Alcohol dependence
17. Chronic narcotic use that cannot be interrupted
18. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
BHB Concentration in blood | 1 Year
  Beta-hydroxybutyrate concentration in blood
Minutes at maximum exertion [Exercise Capacity] | 1 Year
  Minutes at maximum exertion
Left ventricular ejection fraction (%) | 1 Year
  Left ventricular ejection fraction, measured by echocardiogram
Cardiac output (L/min) | 1 Year
  Cardiac output, measured by echocardiogram
Left ventricular end diastolic diameter (LVEDD) (cm) | 1 Year
  LVEDD, measured by echocardiogram
Insulin concentration | 1 Year
  Insulin concentration in blood
Bicarbonate concentration | 1 Year
  Bicarbonate concentration in blood

CONTACTS AND LOCATIONS:
Overall Officials: J. Eduardo Rame, M.D., Principal Investigator — Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: No